CLINICAL TRIAL: NCT07346209
Title: STudy of Real-world Individualized Precision-oncology
Brief Title: Real-world Trial of Individualized Precision Oncology
Acronym: STRIPe
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jason K. Sicklick, M.D., Professor of Surgery and Pharmacology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 813379
Record Dates: First submitted 2026-01-14; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Cancer; Unresectable Carcinoma
Keywords: Precision medicine; Molecularly matched therapy; Tumor molecular alterations; Molecular Tumor Board
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Molecularly matched therapy (Experimental): Molecularly matched therapy based on tumor's molecular profile.
  Interventions: Drug: Molecularly matched therapy
- Standard of care (Active Comparator): Standard of care treatment.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Molecularly matched therapy — Molecularly matched therapy, as identified by a molecular tumor board, to match molecular alterations/biomarkers found in the tumor or circulating tumor DNA.
  Arms: Molecularly matched therapy
Drug: Standard of care — Standard of care therapy for the tumor type.
  Arms: Standard of care

SUMMARY:
The goal of this clinical trial is to learn if drugs that are matched to tumor DNA mutations work to treat metastatic solid cancers in adults. The main questions it aims to answer are:

Is tumor worsening delayed for a longer period of time if patients take drugs that match DNA mutations, compared to if they take standard of care drugs?

Researchers will compare drugs matched to tumor DNA mutations to standard of care drugs to see if the matched drugs work better, and to see if tumor worsening can be delayed for longer the more DNA mutations the drugs target.

Participants will:

Take drugs matched to tumor DNA mutations or standard of care drugs based on the regular dosing schedule of the drugs.

Visit the clinic every approximately 2 months for checkups and tumor imaging.

DETAILED DESCRIPTION:
Next generation sequencing and multi-omic technologies have revealed that advanced or metastatic solid cancers often have complex molecular profiles with multiple driver alterations/biomarkers that are different from patient to patient. This molecular complexity and heterogeneity require customized treatment regimens targeting multiple driving molecular alterations/biomarkers while ensuring patient safety.

The investigators conducted previously a preliminary trial on optimized personalized-precision oncology. Personalized-precision oncology entails matching patients to the best drug(s) for their tumor - including drug combinations never studied before - at the right doses to the right patients. That study demonstrated that therapy matched to each cancer's complex and unique molecular profile, as suggested by an expert molecular tumor board, is feasible and safe. In addition, the investigators showed that receipt of therapy targeting a higher proportion of molecular alterations/biomarkers in the tumor was strongly associated with longer progression free survival.

The present randomized study aims to expand the previous findings to evaluate efficacy and safety of molecularly matched therapy in metastatic unresectable cancers and to develop innovative machine learning models to better predict optimal treatment for validation in future trials.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Aged at least 18 years.
4. Metastatic or unresectable solid cancers (all) with a 2-year cancer-associated mortality of ≥ 50%, or immediate prior progression free survival < 4 months, or life expectancy between 6 and 16 months as determined at prescreening and/or enrollment due to cancer diagnosis.
5. Previous treatment with up to 2 lines of cancer therapy before enrollment.
6. Available results of tumor imaging performed within 4 weeks prior to randomization or eligible to obtain imaging as part of routine care. Note that patients are not eligible if their tumor imaging was performed more than 4 weeks before randomization, or if the imaging to be performed at screening is within 6 weeks of their previous imaging.
7. Measurable disease by RECIST v 1.1 based on computed tomography, magnetic resonance imaging or positron emission tomography/computed tomography scan performed within 4 weeks prior to randomization.
8. Case discussed by Molecular Tumor Board with consensus treatment recommendation(s).
9. Presence of at least 1 tumor-derived molecular alteration/biomarker with a molecularly matched therapy option per Molecular Tumor Board recommendation.

   1. Molecular profile needs to be performed in tumor tissue or circulating tumor DNA collected in the 6 months before enrollment and analyzed by next generation sequencing, immunohistochemistry, and/or alternative technology in a Clinical Laboratory Improvement Amendments-accredited and College of American Pathologists-certified clinical laboratory.
   2. All prior pathology and molecular studies may be reviewed and considered by the Molecular Tumor Board.
   3. Molecularly matched therapy options are restricted to Food and Drug Administration-approved drugs.
10. Eligible for at least 1 additional unmatched standard of care therapy.
11. Eastern Cooperative Oncology Group performance status score of 0 or 1.
12. At the time of the screening/baseline visit, patients must be off prior antibody therapy for at least 3 half-lives, and other anti-tumor agents for at least 5 half-lives, or total 3 weeks from the last day of treatment, whichever is shortest.
13. Adequate hematologic, hepatic, and renal function, as specified below:

    1. Absolute Neutrophil Count ≥ 1.5 x 10^9/L
    2. Hemoglobin ≥ 9 g/dL
    3. Platelets ≥ 50 x 10^9/L
    4. Serum total bilirubin < 2.0 x upper limit of normal
    5. Aspartate aminotransferase and alanine aminotransferase ≤ 5 x upper limit of normal
    6. Serum creatinine ≤ 1.5 x upper limit of normal or calculated creatinine clearance ≥ 50ml/min based upon the Cockcroft-Gault Equation [CrCl = (140-age) * actual weight (in kg) * (0.85 if female) / (72 * Cr)].
14. For participants able to become pregnant or cause a pregnancy: use of highly effective contraception during treatment with the study therapy and for 3 months afterwards.

Exclusion Criteria:

1. Presence of very high tumor mutational burden as ≥ 20 mutations/megabase.
2. Presence of a microsatellite instability-high as defined by the testing laboratory.
3. Deficiency of mismatch repair genes: MLH1, MSH2, MSH6, or PMS2.
4. Molecular Tumor Board treatment recommendation is a monotherapy with an immune checkpoint inhibitor.
5. Molecular Tumor Board treatment recommendation is considered a standard of care regimen per NCCN guidelines (including treatments considered useful in certain circumstances).

   * Example 1: Presence of BRAF V600E in lung cancer as the sole molecularly matched target is ineligible, given Food and Drug Administration approval of combination BRAFi/MEKi.
   * Example 2: Presence of BRAF V600E and CDKN2A mutation in lung cancer is eligible, if the Molecular Tumor Board recommendation is the non-standard of care combination of BRAFi/MEKi + CDK4/6i
   * Example 3: Presence of KRAS G12C in breast cancer is eligible as the use of KRAS inhibitors for this specific tumor type is not standard of care.
   * Example 4: Presence of KRAS G12A mutation in colon cancer is eligible if the Molecular Tumor Board recommendation is for non-standard of care MEKi.
6. Newly diagnosed symptomatic brain metastases requiring immediate treatment. Note that patients with asymptomatic or treated stable brain metastases not requiring steroids can be enrolled.
7. Increase of Eastern Cooperative Oncology Group performance status of ≥ 1 point in the 30 days prior to enrollment.
8. Pregnancy or lactation.
9. Known allergic reactions to components of the therapy.
10. Other conditions that preclude study participation at the discretion of the treating physician (e.g., organ or bone marrow dysfunction).
11. Patient is in hospice care.
12. Two oncologists disagree on prognosis or cancer resectability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2031-03 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 1 year
  Duration of time from randomization until objective tumor progression, clinical progression, treatment discontinuation due to inability to tolerate study therapy, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jason K. Sicklick, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sicklick JK, Kato S, Okamura R, Patel H, Nikanjam M, Fanta PT, Hahn ME, De P, Williams C, Guido J, Solomon BM, McKay RR, Krie A, Boles SG, Ross JS, Lee JJ, Leyland-Jones B, Lippman SM, Kurzrock R. Molecular profiling of advanced malignancies guides first-line N-of-1 treatments in the I-PREDICT treatment-naive study. Genome Med. 2021 Oct 4;13(1):155. doi: 10.1186/s13073-021-00969-w. PMID 34607609
- [Background] Sicklick JK, Kato S, Okamura R, Schwaederle M, Hahn ME, Williams CB, De P, Krie A, Piccioni DE, Miller VA, Ross JS, Benson A, Webster J, Stephens PJ, Lee JJ, Fanta PT, Lippman SM, Leyland-Jones B, Kurzrock R. Molecular profiling of cancer patients enables personalized combination therapy: the I-PREDICT study. Nat Med. 2019 May;25(5):744-750. doi: 10.1038/s41591-019-0407-5. Epub 2019 Apr 22. PMID 31011206
- [Background] Kato S, Kim KH, Lim HJ, Boichard A, Nikanjam M, Weihe E, Kuo DJ, Eskander RN, Goodman A, Galanina N, Fanta PT, Schwab RB, Shatsky R, Plaxe SC, Sharabi A, Stites E, Adashek JJ, Okamura R, Lee S, Lippman SM, Sicklick JK, Kurzrock R. Real-world data from a molecular tumor board demonstrates improved outcomes with a precision N-of-One strategy. Nat Commun. 2020 Oct 2;11(1):4965. doi: 10.1038/s41467-020-18613-3. PMID 33009371